CLINICAL TRIAL: NCT02825004
Title: Recognizing and Preventing Burnout: A Pilot Randomized Controlled Trial
Brief Title: Recognizing and Preventing Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Paolo Banfi, M.D., Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDG_BURN01_HP
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Burnout, Professionals
Keywords: Burnout; Health Care Workers; Coping Skills; Clinical Trial
MeSH Terms: conditions — Burnout, Psychological | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychological Intervention (Experimental): All the professionals workers involved in the experimental group will attend three intensive psychological meetings about emotional exhaustion, depersonalisation, low personal accomplishment and how to improve coping skills.
  Interventions: Behavioral: Psychological Intervention
- Control Group (No Intervention): There is not any intervention.

INTERVENTIONS:
Behavioral: Psychological Intervention
  Arms: Psychological Intervention

SUMMARY:
The purpose of this study is to prevent burnout and offer the hospital staff a space for processing the emotional experiences.

ELIGIBILITY:
Inclusion Criteria:

* Doctors, physiotherapists, nurses and care workers
* Be a Professional Worker at the Rehabilitation Respiratory Unit
* Age > 18 years old

Exclusion Criteria:

* Refusal at the Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes in burnout, as assessed by the Maslach Burnout Inventory (MBI) (Maslach C., 1981) between baseline (T0), 6 months (T1) and 12 months (T2) | At the baseline (T0), 6 months (T1) and 12 months (T2)

SECONDARY OUTCOMES:
Changes in coping strategies as assessed by the Coping Orientation to Problems Experienced (COPE) (Carver et al., 1989) between baseline (T0), 6 months (T1) and 12 months (T2) | At the baseline (T0), 6 months (T1) and 12 months (T2)
Changes in psychological symptoms as assessed by the Symptom Checklist-90-R (Prunas et al., 2012) between baseline (T0), 6 months (T1) and 12 months (T2) | At the baseline (T0), 6 months (T1) and 12 months (T2)

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Banfi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Prunas A, Sarno I, Preti E, Madeddu F, Perugini M. Psychometric properties of the Italian version of the SCL-90-R: a study on a large community sample. Eur Psychiatry. 2012 Nov;27(8):591-7. doi: 10.1016/j.eurpsy.2010.12.006. Epub 2011 Feb 21. PMID 21334861
- [Result] Kleijweg JH, Verbraak MJ, Van Dijk MK. The clinical utility of the Maslach Burnout Inventory in a clinical population. Psychol Assess. 2013 Jun;25(2):435-41. doi: 10.1037/a0031334. Epub 2013 Jan 28. PMID 23356679
- [Result] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629